CLINICAL TRIAL: NCT04213625
Title: Do Patients Perceive Surgeons Who Provide Personal Information ("Self-disclosure") as More Trustworthy and Empathetic?
Brief Title: Do Patients Perceive Surgeons Who Provide Personal Information as More Trustworthy and Empathetic?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Deemed infeasible.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Professor, Dean associate of surgery department, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-06-0047
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Trust

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Information sheet with only their surgeon's educational background.
- Intervention (Experimental): Experimental group will receive an information sheet with their surgeon's educational and personal background.
  Interventions: Other: Surgeon Personal Background

INTERVENTIONS:
Other: Surgeon Personal Background — Experimental group will receive an information sheet with their surgeon's educational and personal background.
  Personal Background
  * Favorite outdoor activity/form of exercise
  * Favorite hobby
  * Family information (children, pets)
  * Single sentence about how the clinician conceptualizes excellent patient care
  Arms: Intervention

SUMMARY:
Prior studies have shown that patient trust in their physician is associated with better health outcomes and lower levels of emotional distress. Patients who have low levels of trust in their physician are less satisfied and less likely to adhere to their physician recommendations. As such, there is a need to better understand factors related to patient trust in their physician.

Purpose: To understand whether patient awareness of a surgeon's personal background improves patient trust in their surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age 18 years or greater) visiting a single orthopaedic hand surgeon
* English fluency and literacy
* Ability to take informed consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Wake Forest -Trust in Physician score | Immediately after the clinic visit, patients are given the survey to complete.
  Before the clinic visit, the research assistant will give patients a sheet that gives them info on their surgeon. Control group will receive an information sheet with only their surgeon's educational background. Experimental group will receive an information sheet with their surgeon's educational and personal background. Immediately after the clinic visit, the research assistant will ask patients to complete Wake Forest Trust in physician survey. Response choices (coding) are: Strongly Agree (5), Agree (4), Neutral (3), Disagree (2), Strongly Disagree (1). Responses are summed (range 5-25) with higher scores indicating more trust.
Jefferson Scale of Perceived Physician Empathy | Immediately after the clinic visit, patients are given the survey to complete.
  Before the clinic visit, the research assistant will give patients a sheet that gives them info on their surgeon. Control group will receive an information sheet with only their surgeon's educational background. Experimental group will receive an information sheet with their surgeon's educational and personal background. Immediately after the clinic visit, the research assistant will ask patients to complete the Jefferson Scale of Patient Perceptions of Physician Empathy. Each item is answered on a 7-point Likert-type scale (from Strongly Disagree = 1 to Strongly Agree = 7), with higher score indicating more empathy.